CLINICAL TRIAL: NCT03188796
Title: The VITDALIZE Study: Effect of High-dose Vitamin D3 on 28-day Mortality in Adult Critically Ill Patients With Severe Vitamin D Deficiency: a Multicenter, Placebo-controlled Double-blind Phase III Randomized Controlled Trial (RCT)
Brief Title: The VITDALIZE Study: Effect of High-dose Vitamin D3 on 28-day Mortality in Adult Critically Ill Patients
Acronym: VITDALIZE
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Medical University of Graz (Other)
Collaborators: Medical University of Vienna (Other); Hospital Barmherzige Brüder St. Veit (Unknown); Klinikum Klagenfurt am Wörthersee (Other); Johannes Kepler University of Linz (Other); Krankenhaus Barmherzige Schwestern Linz (Other); Barmherzige Brüder Vienna (Other); Erasme University Hospital (Other); The Queen Elizabeth Hospital (Other); Goethe University (Other); Kages (Other); KABEG Management (Other); Centre Hospitalier Régional de la Citadelle (Other); Centre Hospitalier Universitaire de Charleroi (Other); Centre Hospitalier Universitaire Mons (Unknown); Wuerzburg University Hospital (Other); Royal Bolton Hospital NHS Foundation Trust (Other); Heartlands Hospital (Unknown); Royal Oldham Hospital (Unknown); East Lancashire Hospitals NHS Trust (Other); University of Plymouth (Other); Royal Victoria Hospital, Belfast (Other); Great Western Hospital (Unknown); Mid Yorkshire Teaching NHS Trust (Other); Musgrove Park Hospital (Unknown); Scunthorpe General Hospital (Unknown); Guy's and St Thomas' NHS Foundation Trust (Other); Nottingham University Hospitals (Unknown); Hospital Barmherzige Brüder Graz (Unknown); University Hospital Kiel (Unknown); University Hospital, Bonn (Other); Johannes Gutenberg University Mainz (Other); University Hospital, Essen (Other); Klinikum rechts der Isar der TUM (Unknown); Landeskrankenhaus Villach (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: VITDALIZE 1.0
Record Dates: First submitted 2017-06-13; First posted 2017-06-15 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-10

CONDITIONS: Critical Illness; Vitamin D Deficiency; Covid19
Keywords: vitamin D; critical care; COVID-19
MeSH Terms: conditions — Critical Illness; Vitamin D Deficiency; COVID-19 | interventions — Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): oral/enteral loading dose of 37.5 ml MCT followed by 10 drops daily for 90 days
  Interventions: Drug: Placebo
- High Dose Vitamin D3 (Experimental): oral/enteral pharmacological dose of cholecalciferol (vitamin D3) - total dose 900,000
  * loading dose of 540,0000 (dissolved in 37.5 ml of medium chain triglycerides - MCT)
  * followed by 4000 IU daily (10 drops) for the entire active study period (90 days)
  Interventions: Drug: Cholecalciferol

INTERVENTIONS:
Drug: Cholecalciferol — oral/enteral loading dose of 37.5 ml MCT including 540,000 IU vitamin D3 followed by 10 drops daily (4000 IU) for 90 days
  Other Names: Vitamin D3
  Arms: High Dose Vitamin D3
Drug: Placebo — oral/enteral loading dose of 37.5 ml MCT followed by 10 drops daily for 90 days
  Arms: Placebo

SUMMARY:
In the VITdAL-ICU trial using a large oral dose of vitamin D3 in 480 adult critically ill patients, there was no benefit regarding the primary endpoint hospital length of stay. However, the predefined subgroup with severe vitamin D deficiency (25(OH)D ≤ 12ng/ml) had significantly lower 28-day mortality (36.3% placebo vs. 20.4% vitamin D group, hazard ratio (HR) 0.52 (0.30-0.89), number needed to treat = 6). Therefore, high-dose vitamin D3 in a population of severely vitamin D deficient critically ill patients is a promising and inexpensive intervention that requires confirmatory multicenter studies.

To date, only 7 interventions (e.g. noninvasive ventilation or prone positioning) have ever demonstrated mortality benefit for Intensive Care Unit (ICU) patients in multicenter trials. In case of benefit, vitamin D treatment in critically ill patients could be immediately implemented worldwide.

DETAILED DESCRIPTION:
A very limited number of intervention trials, most including less than 30 patients, have been published. The only phase III study, our VITdAL-ICU study recruited from 2010 to 2012 and (n=475) did not find a difference in the primary endpoint "length of hospital stay" between placebo and high-dose vitamin D3. However, there was a non-significant absolute risk reduction in all-cause hospital mortality in the total population. The difference was larger (17.5%) and significant in the predefined subgroup of patients with severe vitamin D deficiency at baseline, see Kaplan Meier curve below (n=200, 28.6 vs 46.1%, p=0.01, 0.56 (0.35-0.90) ), corresponding to a number needed to treat of 6. (51) As this was only a secondary endpoint in the predefined subgroup with severe vitamin D deficiency, this finding is hypothesis generating and requires further study, leading to this application.

In our study, we were unable to identify a mechanism by which this benefit was achieved. Interestingly, looking at the causes of death, the vitamin D group seemed to benefit in every category.

The VITDALIZE study is a pragmatic, multicenter, placebo-controlled double-blind randomized controlled phase III trial in adult critically ill patients which will be conducted in academic and non-academic centers. The sponsor is the Medical University of Graz, Austria.

Subjects will be randomised in a 1:1 ratio to receive either of the two treatments:

Vitamin D: oral/enteral pharmacological dose of cholecalciferol (vitamin D3)

* total dose 900,000
* loading dose of 540,0000 (dissolved in 37.5 ml of medium chain triglycerides - MCT) followed by 4000 IU daily (10 drops) for the entire active study period (90 days)

Placebo: identical regime - loading dose of 37.5 ml MCT followed by 10 drops daily

This study uses a group sequential design, with one interim analysis when 50% of the planned enrolled patients in each arm (N=600 per arm) have completed their day 28 assessment by the independent data safety monitoring board. The enrollment of patients will continue while the interim analyses is performed.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years
* Anticipated ICU stay ≥ 48 hours
* Admission to ICU ≤ 72 hours before screening
* Severe vitamin D deficiency (≤12 ng/ml or undetectable)

Exclusion Criteria:

* Severe gastrointestinal dysfunction (> 400 ml residual volume)/unable to take study medication
* Do not resuscitate (DNR) order/imminent death
* hypercalcemia
* known recent nephrolithiasis, active tuberculosis or sarcoidosis
* pregnancy/lactation
* not deemed appropriate by study team/physician

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2400 (Estimated)
Dates: Start 2017-10-10 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
28-day mortality | 28 days
  all-cause mortality

SECONDARY OUTCOMES:
Hospital Length of stay | 90 days
  Length of stay in days
Hypercalcemia at day 5 | Day 5 - 48 hours tolerance
Hospital readmissions | 90 days
  Number of readmissions

CONTACTS AND LOCATIONS:
Overall Officials: Karin Amrein, MD, MSc, Principal Investigator — Medical University of Graz
Locations (18):
- Austria (12):
  - LKH Enzenbach, Enzenbach
  - LKH Feldbach, Feldbach
  - Medical University of Graz, Graz
  - Klinikum am Wörthersee, Klagenfurt
  - LKH Hochsteiermark Standort Leoben, Leoben
  - Barmherzige Schwestern, Linz
  - Kepler Universitätsklinikum Linz, Linz
  - Krankenhaus Schwarzach, Schwarzach im Pongau
  - Barmherzige Brüder, Vienna
  - Kaiser Franz Josef Spital Wien, Vienna
  - Medical University of Vienna, Vienna
  - LKH Villach, Villach
- Belgium (4):
  - Erasme Hospital, Brussels
  - CHU de Charleroi, Charleroi
  - CHR Citadelle, Liège
  - CHU Ambroise Pare, Mons
- University Hospital Wuerzburg, Würzburg, Germany
- University of Birmingham, Birmingham, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Amrein K, Schnedl C, Holl A, Riedl R, Christopher KB, Pachler C, Urbanic Purkart T, Waltensdorfer A, Munch A, Warnkross H, Stojakovic T, Bisping E, Toller W, Smolle KH, Berghold A, Pieber TR, Dobnig H. Effect of high-dose vitamin D3 on hospital length of stay in critically ill patients with vitamin D deficiency: the VITdAL-ICU randomized clinical trial. JAMA. 2014 Oct 15;312(15):1520-30. doi: 10.1001/jama.2014.13204. PMID 25268295
- [Background] Amrein K, Christopher KB, McNally JD. Understanding vitamin D deficiency in intensive care patients. Intensive Care Med. 2015 Nov;41(11):1961-4. doi: 10.1007/s00134-015-3937-4. Epub 2015 Jul 4. No abstract available. PMID 26142054
- [Background] Amrein K. Vitamin D status in critical care: Contributor or marker of poor health? Lung India. 2014 Jul;31(3):299-300. No abstract available. PMID 25125826
- [Background] Amrein K, Papinutti A, Mathew E, Vila G, Parekh D. Vitamin D and critical illness: what endocrinology can learn from intensive care and vice versa. Endocr Connect. 2018 Dec 1;7(12):R304-R315. doi: 10.1530/EC-18-0184. PMID 30352414
- [Background] National Heart, Lung, and Blood Institute PETAL Clinical Trials Network; Ginde AA, Brower RG, Caterino JM, Finck L, Banner-Goodspeed VM, Grissom CK, Hayden D, Hough CL, Hyzy RC, Khan A, Levitt JE, Park PK, Ringwood N, Rivers EP, Self WH, Shapiro NI, Thompson BT, Yealy DM, Talmor D. Early High-Dose Vitamin D3 for Critically Ill, Vitamin D-Deficient Patients. N Engl J Med. 2019 Dec 26;381(26):2529-2540. doi: 10.1056/NEJMoa1911124. Epub 2019 Dec 11. PMID 31826336
- [Background] Kobayashi H, Amrein K, Mahmoud SH, Lasky-Su JA, Christopher KB. Metabolic phenotypes and vitamin D response in the critically ill: A metabolomic cohort study. Clin Nutr. 2024 Nov;43(11):10-19. doi: 10.1016/j.clnu.2024.09.030. Epub 2024 Sep 18. PMID 39307095
- [Background] Geiger C, McNally JD, Christopher KB, Amrein K. Vitamin D in the critically ill - update 2024. Curr Opin Clin Nutr Metab Care. 2024 Nov 1;27(6):515-522. doi: 10.1097/MCO.0000000000001068. Epub 2024 Aug 26. PMID 39302310
- [Derived] Shakoor H, Feehan J, Al Dhaheri AS, Cheikh Ismail L, Ali HI, Alhebshi SH, Apostolopoulos V, Stojanovska L. Role of vitamin D supplementation in aging patients with COVID-19. Maturitas. 2021 Oct;152:63-65. doi: 10.1016/j.maturitas.2021.03.006. Epub 2021 Mar 16. No abstract available. PMID 33757717
- [Derived] Amrein K, Parekh D, Westphal S, Preiser JC, Berghold A, Riedl R, Eller P, Schellongowski P, Thickett D, Meybohm P; VITDALIZE Collaboration Group. Effect of high-dose vitamin D3 on 28-day mortality in adult critically ill patients with severe vitamin D deficiency: a study protocol of a multicentre, placebo-controlled double-blind phase III RCT (the VITDALIZE study). BMJ Open. 2019 Nov 12;9(11):e031083. doi: 10.1136/bmjopen-2019-031083. PMID 31722941